CLINICAL TRIAL: NCT04502264
Title: Effects of EMG-driven Robot-assisted Therapy for the Distal Upper Limb Motor Function in the Chronic Stroke Patients With Botox Injections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: (745)108A-61
Record Dates: First submitted 2020-07-22; First posted 2020-08-06 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Chronic Stroke; Spasticity as Sequela of Stroke; Robotic Rehabilitation
Keywords: Hand of hope; hand robot; Botulinum toxin
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin, hand robot training, occupational therapy (Experimental): Patient would receive Botulinum toxin (Injections of 100~400U of Botox in the upper limb muscle with a 2ml/100U dilution), robot-assisted therapy (Hand of Hope training), and standard occupational therapy.
  Interventions: Device: Hand of Hope; Drug: Botulinum toxin type A injection
- Botulinum toxin, occupational therapy (Active Comparator): Patient would receive Botulinum toxin (Injections of 100~400U of Botox in the upper limb muscle with a 2ml/100U dilution) and standard occupational therapy.
  Interventions: Drug: Botulinum toxin type A injection

INTERVENTIONS:
Device: Hand of Hope — A virtual reality (VR)-based, electromyography (EMG)-driven, and task-oriented hand robot.
  Arms: Botulinum toxin, hand robot training, occupational therapy
Drug: Botulinum toxin type A injection — A safe agent representing the gold standard treatment for focal spasticity.

SUMMARY:
Over fifty percent of stroke patients experience chronic arm hand performance problems, compromising independence in daily life activities and quality of life. Traditionally, the effectiveness of rehabilitation in improving functioning for stroke patients more than 6 months has not been proven. However, spontaneous neurological recovery reaches the plateau at 3~6 months later.

Hand of Hope is a virtual reality (VR)-based, electromyography (EMG)-driven, and task-oriented hand robot. Otherwise, it needs patients to have active participation during the intervention which is critical for motor recovery after stroke. Robotic rehabilitation devices have the potential to deliver high-intensity, reproducible therapy. Robot-assisted task-oriented training had been proposed by several researchers, but the evidence of clinical effectiveness in highly functional chronic stroke patients is still lack.

Spasticity is a common disorder which occurs following stroke. The prevalence of post-stroke spasticity can be as high as 46% in the chronic phase (over 3 months). Spasticity impacted activities of daily living, quality of life, pain, and functional impairments. Long-term spasticity may lead to tendon contracture and limb deformities. Botulinum toxin injection, which mostly used in chronic phase (over 6 months), had been proved to be a safe agent representing the gold standard treatment for focal spasticity, while avoiding systemic effects. But the effects of botulism toxin on functional ability are still unclear. Moreover, there is insufficient evidence on adjunctive therapies following botulism toxin.

The purpose of the present study is to examine the effects of botulinum toxin injection combined with Hand of Hope and standard occupational therapy on upper extremity function, and compares the findings to those of amount-matched chronic stroke survivors who received only Botulinum toxin injection and standard occupational therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20-85 year-old
* The onset of stroke must be at least 6 month previously
* The stroke must be the first event
* The stroke must be unilateral brain lesion
* Spasticity measured as Modified Ashworth scale during 1+ to 3
* Score at least 1 point in the wrist subtest of Fugl-Meyer Assessment
* Brunnstrom stage of proximal upper limb at least 3, distal upper limb between 2 to 5
* No impairment in visual tracking ability
* No impairment in proprioception

Exclusion Criteria:

* Severe joints pain of hand or finger at affected limb
* Fracture of affected limb in three months
* Brunnstrom stage of proximal upper limb not more than 2, distal upper limb more than 5

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
modified Ashworth scale | 14 weeks
  Modified Ashworth scale is a scale for spasticity evaluation, while 0 means no spasticity, 1 means slight increase in muscle tone, 1+ means more muscle tone than score equels 1, 2 means more marked muscle tone, 3 means passive movement is difficult, and 4 means rigidity. We would record modified Ashworth scale at upper limb of the hemiplegic patients.
H-reflex | 14 weeks
  H-reflex is a method of electricophysilogic evaluation for spasticity in nerve conduction study, while decreased latency means stronger muscle tone and prolonged latency means weaker muscle tone. H-reflex of all limbs at these patients would be recorded.
Box & Block Test | 14 weeks
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. 150 blocks is set up at the test box, and clients are scored based on the number of blocks transferred from one compartment to the other compartment in 60 seconds. Higher scores are indicative of better manual dexterity.
Nine Hole Peg Test | 14 weeks
  The Nine-Hole Peg Test is used to measure finger dexterity by asking the client to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible. Scores are based on the time taken to complete the test activity, recorded in seconds.
World Health Organization Quality of Life (WHOQOL-BREF)-Taiwan version | 14 weeks
  The World Health Organization Quality of Life (WHOQOL-BREF) is a 28-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (4 items), and environmental health (9 items); with another 2 items about general condition and overall quality of life. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. The higher scores equals better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng-Hsin general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided